CLINICAL TRIAL: NCT03190941
Title: A Phase I/II Study Administering Peripheral Blood Lymphocytes Transduced With a Murine T-Cell Receptor Recognizing the G12V Variant of Mutated RAS in HLA-A*11:01 Patients
Brief Title: Administering Peripheral Blood Lymphocytes Transduced With a Murine T-Cell Receptor Recognizing the G12V Variant of Mutated RAS in HLA-A*11:01 Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 170113; 17-C-0113
Record Dates: First submitted 2017-06-16; First posted 2017-06-19 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11-26

CONDITIONS: Pancreatic Cancer; Gastric Cancer; Gastrointestinal Cancer; Colon Cancer; Rectal Cancer
Keywords: KRAS; HRAS; NRAS; Cell Therapy; Immunotherapy
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms; Gastrointestinal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cyclophosphamide; fludarabine; aldesleukin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Phase I (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + escalating doses of anti-KRAS G12V mTCR PBL + high-dose aldesleukin
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Anti-KRAS G12V mTCR PBL; Drug: Aldesleukin
- 2/Phase II (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + MTD of anti-KRAS G12V mTCR PBL + high-dose aldesleukin
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Anti-KRAS G12V mTCR PBL; Drug: Aldesleukin

INTERVENTIONS:
Drug: Cyclophosphamide — Days -7 and -6: Cyclophosphamide 60 mg/kg/day x 2 days IV in 250 mL D5W infused simultaneously with mesna 15 mg/kg/day over 1 hour x 2 days.
Drug: Fludarabine — Days -7 to -3: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days.
Biological: Anti-KRAS G12V mTCR PBL — Day 0: Cells will be infused intravenously on the Patient Care Unit over 20-30 minutes (2-4 days after the last dose of fludarabine).
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg IV (based on total body weight) over 15 minutes approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to 3 days (maximum 9 doses).

SUMMARY:
Background:

A new cancer therapy involves taking white blood cells from a person, growing them in the lab, genetically modifying them, then giving them back to the person. This therapy is called gene transfer using anti-KRAS G12V mTCR cells.

Objective:

To see if anti-KRAS G12 V mTCR cells are safe and can shrink tumors.

Eligibility:

Adults at least 18 years old with cancer that has the KRAS G12V molecule on the surface of tumors.

Design:

In another protocol, participants will:

Be screened

Have cells harvested and grown

Have leukapheresis

In this protocol, participants will have the procedures below.

Participants will be admitted to the hospital.

Over 5 days, participants will get 2 chemotherapy medicines as an infusion via catheter in the upper chest.

A few days later, participants will get the anti-KRAS G12V mTCR cells via catheter.

For up to 3 days, participants will get a drug to make the cells active.

A day after getting the cells, participants will get a drug to increase their white blood cell count. This will be a shot or injection under the skin.

Participants will recover in the hospital for 1-2 weeks. They will have lab and blood tests.

Participants will take an antibiotic for at least 6 months.

Participants will have visits every few months for 2 years, and then as determined by their doctor.

Visits will be 1-2 days. They will include lab tests, imaging studies, and physical exam. Some visits may include leukapheresis or blood drawn.

Participants will have blood collected over several years.

DETAILED DESCRIPTION:
Background:

* We generated an HLA-A*11:01-restricted murine T-cell receptor (mTCR) that specifically recognizes the G12V-mutated variant of KRAS (and other RAS family genes), expressed by many human cancers and constructed a single retroviral vector that contains alpha and beta chains that confer recognition of this antigen when transduced into PBL.
* In co-cultures with HLA-A*11:01+ target cells expressing this mutated oncogene, mTCR transduced T cells lyse target cells and secrete IFN-gamma with high specificity.

Objectives:

Primary objectives:

* Phase I: Determine the safety of administering PBL transduced with anti-KRAS G12V mTCR in concert with preparative lymphodepletion and high-dose interleukin-2 (IL-2; aldesleukin).
* Phase II: Determine if anti-KRAS G12V mTCR-transduced PBL can mediate the regression of tumors harboring the RAS G12V mutation.

Eligibility:

Patients must be/have:

* Age greater than or equal to 18 years and less than or equal to 72 years
* HLA-A*11:01 positive
* Metastatic or unresectable RAS G12V-expressing cancer which has progressed after standard therapy (if available).

Patients may not have:

-Allergies or hypersensitivities to high-dose aldesleukin, cyclophosphamide or fludarabine.

Design:

* This is a Phase I/II, single center study of PBL transduced with anti-KRAS G12V mTCR in HLA-A*11:01 positive patients with advanced solid tumors expressing G12V mutated RAS.
* PBMC obtained by leukapheresis will be cultured in the presence of anti-CD3 (OKT3) and aldesleukin in order to stimulate T-cell growth.
* Transduction is initiated by exposure of these cells to retroviral vector supernatant containing replication-incompetent virus encoding the anti-KRAS G12V mTCR.
* All patients will receive a non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine.
* On day 0, patients will receive their PBL transduced with the anti-KRAS G12V mTCR and will then begin high-dose aldesleukin.
* A complete evaluation of lesions will be conducted approximately 6 weeks (+/- 2 weeks) after treatment.
* The study will be conducted using a phase I/II Simon minimax design, with two separate

cohorts for the Phase II component: Cohort 2a, patients with RAS G12V pancreatic

cancer, and Cohort 2b, patients with RAS G12V non-pancreatic cancer.

-A total of up to 110 patients may be required; approximately 24 patients in the phase I portion of the study and 86 (41, plus an allowance of up to 2 non-evaluable per phase II cohort) patients in the phase II portion of the study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Measurable (per RECIST V1.1 criteria, metastatic, or unresectable malignancy expressing G12V mutated KRAS as assessed by one of the following methods: RT-PCR on tumor tissue, tumor DNA sequencing, or any other CLIA-certified laboratory test on resected tissue. Patients shown to have tumors expressing G12V mutated NRAS and HRAS will also be eligible as these oncogenes share complete amino acid homology with G12V mutated KRAS for their first 80 N-terminal amino acids, completely encompassing the target epitope.
* Patients must be HLA-A*11:01 positive as confirmed by the NIH Department of Transfusion Medicine.
* Confirmation of the diagnosis of cancer by the NCI Laboratory of Pathology.
* Patients must have:

  * previously received standard systemic therapy for their advanced cancer and have been either non-responders or have recurred, specifically:

    * Patients with metastatic colorectal cancer must have had at least two systemic chemotherapy regimens that include 5FU, leucovorin, bevacizumab, oxaliplatin, and irinotecan (or similar agents), or have contraindications to receiving those medications.
    * Patients with pancreatic cancer must have received gemcitabine, 5FU, and oxaliplatin (or similar agents), or have contraindications to receiving those medications.
    * Patients with non-small cell lung cancer (NSCLC) must have had appropriate targeted therapy as indicated by abnormalities in ALK, EGFR, or expression of PDL- 1. Other patients must have had platinum-based chemotherapy.
    * Patients with ovarian cancer or prostate cancer must have had approved first-line chemotherapy.

OR

* declined standard treatment
* Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for one month after treatment for the patient to be eligible. Patients

with surgically resected brain metastases are eligible.

* Age greater than or equal to 18 years and less than or equal to 72 years.
* Clinical performance status of ECOG 0 or 1
* Patients must be willing to practice birth control from the time of enrollment on this study and 12 months after the last dose of combined chemotherapy for women and for 4 months after treatment for men.
* Women of child-bearing potential must be willing to undergo pregnancy testing prior to the start of treatment because of the potentially dangerous effects of the treatment on the fetus.

NOTE: Certain malignancies may secrete hormones that produce false positive pregnancy tests. Serial blood testing (e.g. HCG measurements) and/ or ultrasound may be performed for clarification.

* Serology

  * Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive may have decreased immune-competence and thus may be less responsive to the experimental treatment and more susceptible to its toxicities.)
  * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
* Hematology

  * ANC greater than 1000/mm^3 without the support of filgrastim
  * WBC greater than or equal to 2500/mm^3
  * Platelet count greater than or equal to 80,000/mm^3
  * Hemoglobin > 8.0 g/dL. Subjects may be transfused to reach this cut-off.
* Chemistry

  * Serum ALT/AST less than or equal to 5.0 times ULN
  * Total bilirubin less than or equal to 2.0 mg/dL, except in patients with Gilbert s Syndrome, who must have a total bilirubin less than 3.0 mg/dL.
* Patients must have either an eGFR > 60 mL/m (based on serum creatinine and lab nomogram) or a formal 6-24h CrCl > 60 mL/m.
* Patients must have completed any prior systemic therapy at the time of enrollment.

Note: Patients may have undergone minor surgical procedures or limited field radiotherapy within the four weeks prior to enrollment, as long as related major organ toxicities have recovered to less than or equal to grade 1.

* Ability of subject to understand and the willingness to sign a written informed consent document.
* Willing to sign a durable power of attorney.
* Subjects must be co-enrolled on protocol 03C0277.

EXCLUSION CRITERIA:

* Large volume pulmonary irradiation.
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
* Concurrent systemic steroid therapy.
* Active systemic infections requiring anti-infective treatment, coagulation disorders, or any other active or uncompensated major medical illnesses.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune-competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
* History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, or aldesleukin.
* History of coronary revascularization or ischemic symptoms
* For select patients with a clinical history prompting cardiac evaluation: last known LVEF less than or equal to 45%.
* For select patients with a clinical history prompting pulmonary evaluation: known FEV1 less than or equal to 50% or DLCO less than 60%.
* Patients who are receiving any other investigational agents.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2017-09-21 (Actual); Primary Completion 2027-06-29 (Estimated); Study Completion 2028-06-29 (Estimated)

PRIMARY OUTCOMES:
Response rate | 6 weeks and 12 weeks following administration of the cell product, then every 3 months x3, then every 6 months x 2 years, then per PI discretion
  Percentage of patients who have a clinical response (PR+CR) to treatment (objective tumor regression)
Frequency and severity of treatment-related adverse events | From time of cell infusion to two weeks after cell infusion
  Grade and type of toxicity per dose level; fraction of patients who experience a DLT at a given dose level, and number and grade of each type of DLT

CONTACTS AND LOCATIONS:
Overall Officials: James C Yang, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Davis JL, Theoret MR, Zheng Z, Lamers CH, Rosenberg SA, Morgan RA. Development of human anti-murine T-cell receptor antibodies in both responding and nonresponding patients enrolled in TCR gene therapy trials. Clin Cancer Res. 2010 Dec 1;16(23):5852-61. doi: 10.1158/1078-0432.CCR-10-1280. PMID 21138872
- [Background] Wang QJ, Yu Z, Griffith K, Hanada K, Restifo NP, Yang JC. Identification of T-cell Receptors Targeting KRAS-Mutated Human Tumors. Cancer Immunol Res. 2016 Mar;4(3):204-14. doi: 10.1158/2326-6066.CIR-15-0188. Epub 2015 Dec 23. PMID 26701267
- [Background] Abrams SI, Khleif SN, Bergmann-Leitner ES, Kantor JA, Chung Y, Hamilton JM, Schlom J. Generation of stable CD4+ and CD8+ T cell lines from patients immunized with ras oncogene-derived peptides reflecting codon 12 mutations. Cell Immunol. 1997 Dec 15;182(2):137-51. doi: 10.1006/cimm.1997.1224. PMID 9514698
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-C-0113.html